CLINICAL TRIAL: NCT04732871
Title: A Phase 3, Randomized, Open-label, Multi-country Study to Evaluate the Immunogenicity, Safety, Reactogenicity and Persistence of a Single Dose of the RSVPreF3 OA Investigational Vaccine and Different Revaccination Schedules in Adults Aged 60 Years and Above
Brief Title: Immunogenicity, Safety, Reactogenicity and Persistence of an Investigational Respiratory Syncytial Virus (RSV) Vaccine in Adults Aged 60 Years and Above
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 212496; 2024-512291-34 (EudraCT Number)
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Vaccine; Safety; Reactogenicity; Immunogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Masking Description: Open-label study. Both investigator and participant know the identity of the intervention assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RSV_annual Group (Experimental): Participants receive one dose of RSVPreF3 OA investigational vaccine at Day 1 and 2 revaccination doses at 12 months post-Dose 1 and at 24 months post-Dose 1, respectively and are followed up until Month 60.
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- RSV_Flexible revaccination Group (Experimental): Participants receive one dose of RSVPreF3 OA investigational vaccine at Day 1 and 2 revaccination doses at 24 months post-Dose 1 and at 48 months post-Dose 1, respectively and are followed up until Month 60.
  Interventions: Biological: RSVPreF3 OA investigational vaccine
- RSV_1dose Group (Experimental): Participants receive one dose of RSVPreF3 OA investigational vaccine at Day 1 and are followed up until Month 36. At Month 36, participants in this group will be re-randomized in 2 groups: RSV_1dose_M36 (which will receive 1 additional revaccination dose at Month 36 and will be followed up until Month 60) and RSV_1dose_Flexible (which will receive 1 additional revaccination dose at Month 60, and will be followed up until study end at Month 72).
  Interventions: Biological: RSVPreF3 OA investigational vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — RSVPreF3 OA investigational vaccine administered intramuscularly in the deltoid region of the non-dominant arm.

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity, immunogenicity and long-term persistence of immune response up to 5 years following a single dose vaccination of GSK's investigational vaccine RSVPreF3 OA, in adults aged 60 years and above. The study will also evaluate the immunogenicity, safety and reactogenicity of additional vaccine doses given according to different revaccination schedules.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥60 YOA at first vaccination, who live in the community (CD participants) or in a Long-term care facility (LTCF participants).
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed informed consent obtained from the participant prior to performance of any study specific procedure.
* Participants who are medically stable in the opinion of the investigator at the time of first vaccination. Patients with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Serious or unstable chronic illness.
* Recurrent or un-controlled neurological disorders or seizures. Participants with medically-controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study vaccine during the period beginning 30 days before the first dose of study vaccine, or planned use during the study period.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after each dose of study vaccine administration, with the exception of inactivated, split virion and subunit influenza vaccines which can be administered up to 14 days before or from 14 days after each study vaccination.
* Previous vaccination with an RSV vaccine.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the first dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first vaccine dose or planned administration during the study period. For corticosteroids, this will mean prednisone >=20 mg/day, or equivalent. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.

Other exclusions

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Bedridden participants.
* Planned move during the study period that will prohibit participation in the trial until the study end. This includes:
* Planned move during the study period to another LTCF that will prohibit participation in the trial until study end.
* Planned move from the community to a LTCF that will prohibit participation in the trial until study end.
* Participation of any study personnel or their immediate dependants, family, or household members.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1720 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2027-02-15 (Estimated)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (18):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, The Villages, Florida
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Richfield, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Wenatchee, Washington
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Germany (7):
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Goch
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, München
  - GSK Investigational Site, Wallerfing
  - GSK Investigational Site, Würzburg
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Tokyo
- Taiwan (4):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Background] Schwarz TF, Hwang SJ, Ylisastigui P, Liu CS, Takazawa K, Yono M, Ervin JE, Andrews CP, Fogarty C, Eckermann T, Collete D, de Heusch M, De Schrevel N, Salaun B, Lambert A, Marechal C, Olivier A, Nakanwagi P, Lievens M, Hulstrom V. Immunogenicity and Safety Following 1 Dose of AS01E-Adjuvanted Respiratory Syncytial Virus Prefusion F Protein Vaccine in Older Adults: A Phase 3 Trial. J Infect Dis. 2024 Jul 25;230(1):e102-e110. doi: 10.1093/infdis/jiad546. PMID 39052726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The demography, immunogenicity, reactogenicity and safety data currently presented is reported only for the first 12 months of the study timeline. The follow-up data (up to 36 months) will be updated during final posting.
Pre-assignment Details: Out of 1720 participants enrolled in the study, 1653 participants received the study vaccination and were included in the Exposed Set.
Groups:
- RSV_annual: Participants received one dose of RSVPreF3 OA investigational vaccine at Day 1 and 2 revaccination doses at 12 months post-Dose 1 and at 24 months post-Dose 1, respectively and were followed up until the study end (Month 36).
- RSV_flexible Revaccination: Participants received one dose of RSVPreF3 OA investigational vaccine at Day 1 and 1 revaccination dose at 24 months post-Dose 1 and were followed up until the study end (Month 36).
- RSV_1dose: Participants received one dose of RSVPreF3 OA investigational vaccine at Day 1 and were followed up until the study end (Month 36).
Period: Overall Study
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Started | 993 | 329 | 331
Completed | 938 | 317 | 317
Not Completed | 55 | 12 | 14
Not completed — Adverse event (AE) requiring expedited reporting | 9 | 1 | 3
Not completed — Lost to Follow-up | 7 | 4 | 3
Not completed — Consent withdrawal, not due to a serious adverse event (SAE) | 26 | 7 | 6
Not completed — Migrated / moved from the study area | 5 | 0 | 0
Not completed — Other | 1 | 0 | 1
Not completed — Ongoing | 6 | 0 | 1
Not completed — Unsolicited non-serious adverse event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose | Total
Number analyzed (Participants) | 993 | 329 | 331 | 1653
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 70.1 (6.6) | 69.9 (6.7) | 69.9 (6.7) | 70.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 542 | 182 | 180 | 904
  Male | 451 | 147 | 151 | 749
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 2 | 0 | 0 | 2
  Asian | 296 | 102 | 98 | 496
  Black Or African American | 19 | 8 | 6 | 33
  Other - Unspecified | 0 | 0 | 1 | 1
  White | 676 | 219 | 226 | 1121

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response in Terms of Respiratory Syncytial Virus (RSV)-A Neutralizing Antibody Geometric Mean Titers (GMTs) at Day 1
Description: RSV-A neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Day 1
Population: Analysis was performed on the per-protocol (PP)-humoral immunity (HI) set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of humoral immunity at Day 1 and for whom immunogenicity results were available for the specified assay, minus participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 342 | 321 | 319
Titers (ED60) | 832.4 [763.4 to 907.7] | 864.9 [790.6 to 946.1] | 896.8 [815.9 to 985.8]

2. Primary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Day 31
Description: RSV-A neutralizing antibodies were given as GMTs and expressed as ED60.
Time Frame: At Day 31
Population: Analysis was performed on the PP-HI set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of humoral immunity at Day 31 and for whom immunogenicity results were available for the specified assay, minus participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 328 | 300 | 309
Titers (ED60) | 8827.2 [7905 to 9857] | 8906.6 [7972.3 to 9950.3] | 9585.6 [8448.8 to 10875.5]

3. Primary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Month 6
Description: RSV-A neutralizing antibodies were given as GMTs and expressed as ED60.
Time Frame: At Month 6
Population: Analysis was performed on the PP-HI set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of humoral immunity at Month 6 and for whom immunogenicity results were available for the specified assay, minus participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 319 | 294 | 311
Titers (ED60) | 3465.2 [3140.9 to 3823] | 3600.1 [3242.2 to 3997.5] | 4223.1 [3795.3 to 4699]

4. Primary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Month 12
Description: RSV-A neutralizing antibodies were given as GMTs and expressed as ED60.
Time Frame: At Month 12
Population: Analysis was performed on the PP-HI set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of humoral immunity at Month 12 and for whom immunogenicity results were available for the specified assay, minus participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 284 | 291 | 296
Titers (ED60) | 2529.9 [2274.5 to 2814] | 2695.7 [2421.4 to 3001] | 2800.1 [2501.6 to 3134.3]

5. Primary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Day 1
Description: RSV-B neutralizing antibodies measured as GMTs and expressed as ED60.
Time Frame: At Day 1
Population: Analysis was performed on the PP-HI set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of humoral immunity at Day 1 and for whom immunogenicity results were available for the specified assay, minus participants with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 342 | 321 | 320
Titers (ED60) | 1138.7 [1046.2 to 1239.3] | 1325.9 [1206.9 to 1456.6] | 1258.7 [1142 to 1387.4]

6. Primary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Day 31
Description: RSV-B neutralizing antibodies measured as GMTs and expressed as ED60.
Time Frame: At Day 31
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 328 | 300 | 309
Titers (ED60) | 9219.7 [8368.7 to 10157.3] | 9955.2 [9002.1 to 11009.3] | 9756.1 [8785.4 to 10834]

7. Primary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Month 6
Description: RSV-B neutralizing antibodies measured as GMTs and expressed as ED60.
Time Frame: At Month 6
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 319 | 294 | 311
Titers (ED60) | 3886.4 [3563.5 to 4238.6] | 4484.6 [4063.8 to 4949] | 4570.6 [4152 to 5031.4]

8. Primary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Month 12
Description: RSV-B neutralizing antibodies measured as GMTs and expressed as ED60.
Time Frame: At Month 12
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 284 | 291 | 296
Titers (ED60) | 2671.4 [2433.3 to 2932.9] | 3015.4 [2737.9 to 3321] | 2977.1 [2669.6 to 3320]

9. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 Immunoglobulin G (IgG) Antibody Geometric Mean Concentrations (GMCs) at Day 1
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 are performed by enzyme-linked immunosorbent assay (ELISA). The corresponding antibody GMC was expressed in Elisa Laboratory Units/milliliter (ELU/mL).
Time Frame: At Day 1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 342 | 320 | 320
ELU/mL | 7334.7 [6868.3 to 7832.8] | 7437.1 [6948.6 to 7959.9] | 7759 [7212.5 to 8346.8]

10. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Day 31
Description: Serological assays for the determination of IgG antibodies against RSV PreF3 are performed by ELISA. The corresponding antibody GMC was expressed in ELU/mL.
Time Frame: At Day 31
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 328 | 300 | 309
ELU/mL | 86929.7 [80662.7 to 93683.6] | 92664.7 [86050.1 to 99787.8] | 94249.4 [87660.7 to 101333.3]

11. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Month 6
Description: as for outcome 10
Time Frame: At Month 6
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 319 | 294 | 311
ELU/mL | 33855.9 [31405.3 to 36497.7] | 35193.5 [32623.6 to 37965.9] | 36525.7 [33938 to 39310.7]

12. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Month 12
Description: as for outcome 10
Time Frame: At Month 12
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 284 | 291 | 296
ELU/mL | 24733.5 [22994.3 to 26604.2] | 26484.1 [24651.7 to 28452.8] | 27360.3 [25476.7 to 29383]

13. Secondary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Month 18
Description: Month 18 data will be disclosed during final posting. RSV-A neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 18
Reporting Status: Not Posted, anticipated posting 2027-05

14. Secondary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Month 24
Description: Month 24 data will be disclosed during final posting. RSV-A neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 24
Reporting Status: Not Posted, anticipated posting 2027-05

15. Secondary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Month 30
Description: Month 30 data will be disclosed during final posting. RSV-A neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 30
Reporting Status: Not Posted, anticipated posting 2027-05

16. Secondary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Month 36
Description: Month 36 data will be disclosed during final posting. RSV-A neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 36
Reporting Status: Not Posted, anticipated posting 2027-05

17. Secondary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Month 13
Description: Month 13 data will be disclosed during final posting. RSV-A neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 13
Reporting Status: Not Posted, anticipated posting 2027-05

18. Secondary Outcome: Humoral Immune Response in Terms of RSV-A Neutralizing Antibody GMTs at Month 25
Description: Month 25 data will be disclosed during final posting. RSV-A neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 25
Reporting Status: Not Posted, anticipated posting 2027-05

19. Secondary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Month 18
Description: Month 18 data will be disclosed during final posting. RSV-B neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 18
Reporting Status: Not Posted, anticipated posting 2027-05

20. Secondary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Month 24
Description: Month 24 data will be disclosed during final posting. RSV-B neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 24
Reporting Status: Not Posted, anticipated posting 2027-05

21. Secondary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Month 30
Description: Month 30 data will be disclosed during final posting. RSV-B neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 30
Reporting Status: Not Posted, anticipated posting 2027-05

22. Secondary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Month 36
Description: Month 36 data will be disclosed during final posting. RSV-B neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 36
Reporting Status: Not Posted, anticipated posting 2027-05

23. Secondary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Month 13
Description: Month 13 data will be disclosed during final posting. RSV-B neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 13
Reporting Status: Not Posted, anticipated posting 2027-05

24. Secondary Outcome: Humoral Immune Response in Terms of RSV-B Neutralizing Antibody Titers at Month 25
Description: Month 25 data will be disclosed during final posting. RSV-B neutralizing antibodies were given as GMTs and expressed as Estimated Dose: serum dilution giving a 60% reduction of the RSV plaques compared to a control without serum (ED60).
Time Frame: At Month 25
Reporting Status: Not Posted, anticipated posting 2027-05

25. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Month 18
Description: Month 18 data will be disclosed during final posting. Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody GMC was expressed in ELU/mL.
Time Frame: At Month 18
Reporting Status: Not Posted, anticipated posting 2027-05

26. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Month 24
Description: Month 24 data will be disclosed during final posting. Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody GMC was expressed in ELU/mL.
Time Frame: At Month 24
Reporting Status: Not Posted, anticipated posting 2027-05

27. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Month 30
Description: Month 30 data will be disclosed during final posting. Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody GMC was expressed in ELU/mL.
Time Frame: At Month 30
Reporting Status: Not Posted, anticipated posting 2027-05

28. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Month 36
Description: Month 36 data will be disclosed during final posting. Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody GMC was expressed in ELU/mL.
Time Frame: At Month 36
Reporting Status: Not Posted, anticipated posting 2027-05

29. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Month 13
Description: Month 13 data will be disclosed during final posting. Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody GMC was expressed in ELU/mL.
Time Frame: At Month 13
Reporting Status: Not Posted, anticipated posting 2027-05

30. Secondary Outcome: Humoral Immune Response in Terms of RSVPreF3 IgG Antibody GMCs at Month 25
Description: Month 25 data will be disclosed during final posting. Serological assays for the determination of IgG antibodies against RSV PreF3 were performed by ELISA. The corresponding antibody GMC was expressed in ELU/mL.
Time Frame: At Month 25
Reporting Status: Not Posted, anticipated posting 2027-05

31. Secondary Outcome: Cell-Mediated Immunity (CMI) Response in Terms of Frequency of RSVPreF3-specific Cluster of Differentiation CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Day 1
Description: Among markers expressed were interleukin-2/13/17 (IL2, IL13, IL17), cluster of 40 ligand (CD40L), 41BB, tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At Day 1
Population: Analysis was performed on the PP-CMI set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of CMI at Day 1, minus participants with protocol deviations that lead to exclusion.
Measure: Median (Inter-Quartile Range); unit: CD4 atl2_7m/ million of CD4+ cells
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 287 | 93 | 95
CD4 atl2_7m/ million of CD4+ cells | 202 [83 to 376] | 143 [26 to 294] | 171 [65 to 385]

32. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Day 1
Description: Among markers expressed were IL2, IL13, IL17, CD40L, 41BB, TNF α and IFN γ, in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At Day 1
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: CD8 atl2_7m/ million of CD8+ cells
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 287 | 93 | 95
CD8 atl2_7m/ million of CD8+ cells | 33 [1 to 110] | 32 [1 to 103] | 2 [1 to 107]

33. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Day 31
Description: as for outcome 32
Time Frame: At Day 31
Population: Analysis was performed on the PP-CMI set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of CMI at Day 31, minus participants with protocol deviations that lead to exclusion.
Measure: Median (Inter-Quartile Range); unit: CD4 atl2_7m/ million of CD4+ cells
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 245 | 81 | 84
CD4 atl2_7m/ million of CD4+ cells | 1310 [813 to 2155] | 1292.5 [820.5 to 2254] | 1570 [876 to 1971]

34. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Day 31
Description: as for outcome 32
Time Frame: At Day 31
Population: as for outcome 33
Measure: Median (Inter-Quartile Range); unit: CD8 atl2_7m/ million of CD8+ cells
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 245 | 81 | 84
CD8 atl2_7m/ million of CD8+ cells | 26 [1 to 129] | 58 [1 to 143] | 5 [1 to 101]

35. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 6
Description: as for outcome 32
Time Frame: At Month 6
Population: Analysis was performed on the PP-CMI set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of CMI at Month 6, minus participants with protocol deviations that lead to exclusion.
Measure: Median (Inter-Quartile Range); unit: CD4 atl2_7m/ million of CD4+ cells
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 263 | 87 | 86
CD4 atl2_7m/ million of CD4+ cells | 662 [428 to 1026] | 644 [442 to 1100] | 695 [427 to 1131]

36. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 6
Description: as for outcome 32
Time Frame: At Month 6
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: CD8 atl2_7m/ million of CD8+ cells
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 248 | 88 | 85
CD8 atl2_7m/ million of CD8+ cells | 38 [1 to 113] | 24.5 [1 to 103.5] | 26 [1 to 87]

37. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 12
Description: as for outcome 32
Time Frame: At Month 12
Population: Analysis was performed on the PP-CMI set, which included participants from the RSV_annual Group, the RSV_flexible revaccination Group and the RSV_1dose Group who had blood samples collected for testing of CMI at Month 12, minus participants with protocol deviations that lead to exclusion.
Measure: Median (Inter-Quartile Range); unit: CD4 atl2_7m/ million of CD4+ cells
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 257 | 94 | 92
CD4 atl2_7m/ million of CD4+ cells | 564 [348 to 898] | 525 [345 to 818] | 671 [374.5 to 1072.5]

38. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 12
Description: as for outcome 32
Time Frame: At Month 12
Population: as for outcome 37
Measure: Median (Inter-Quartile Range); unit: CD8 atl2_7m/ million of CD8+ cells
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 257 | 94 | 92
CD8 atl2_7m/ million of CD8+ cells | 1 [1 to 81] | 18 [1 to 108] | 22 [1 to 104]

39. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 18
Description: Month 18 data will be disclosed during final posting. Among markers expressed were interleukin-2/13/17 (IL2, IL13, IL17), cluster of 40 ligand (CD40L), 41BB, tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At Month 18
Reporting Status: Not Posted, anticipated posting 2027-05

40. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 18
Description: as for outcome 39
Time Frame: At Month 18
Reporting Status: Not Posted, anticipated posting 2027-05

41. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 24
Description: Month 24 data will be disclosed during final posting. Among markers expressed were interleukin-2/13/17 (IL2, IL13, IL17), cluster of 40 ligand (CD40L), 41BB, tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At Month 24
Reporting Status: Not Posted, anticipated posting 2027-05

42. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 24
Description: as for outcome 41
Time Frame: At Month 24
Reporting Status: Not Posted, anticipated posting 2027-05

43. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 30
Description: Month 30 data will be disclosed during final posting. Among markers expressed were interleukin-2/13/17 (IL2, IL13, IL17), cluster of 40 ligand (CD40L), 41BB, tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At Month 30
Reporting Status: Not Posted, anticipated posting 2027-05

44. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 30
Description: as for outcome 43
Time Frame: At Month 30
Reporting Status: Not Posted, anticipated posting 2027-05

45. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 36
Description: Month 36 data will be disclosed during final posting. Among markers expressed were interleukin-2/13/17 (IL2, IL13, IL17), cluster of 40 ligand (CD40L), 41BB, tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At Month 36
Reporting Status: Not Posted, anticipated posting 2027-05

46. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 36
Description: as for outcome 45
Time Frame: At Month 36
Reporting Status: Not Posted, anticipated posting 2027-05

47. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 13
Description: Month 13 data will be disclosed during final posting. Among markers expressed were interleukin-2/13/17 (IL2, IL13, IL17), cluster of 40 ligand (CD40L), 41BB, tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At Month 13
Reporting Status: Not Posted, anticipated posting 2027-05

48. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 13
Description: as for outcome 47
Time Frame: At Month 13
Reporting Status: Not Posted, anticipated posting 2027-05

49. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD4 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 25
Description: Month 25 data will be disclosed during final posting. Among markers expressed were interleukin-2/13/17 (IL2, IL13, IL17), cluster of 40 ligand (CD40L), 41BB, tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations.
Time Frame: At Month 25
Reporting Status: Not Posted, anticipated posting 2027-05

50. Secondary Outcome: CMI Response in Terms of Frequency of RSVPreF3-specific CD8 atl2_7m T Cells Expressing at Least 2 Activation Markers at Month 25
Description: as for outcome 49
Time Frame: At Month 25
Reporting Status: Not Posted, anticipated posting 2027-05

51. Secondary Outcome: Number of Participants With at Least One Solicited Administration-site Event Following Vaccination at Day 1
Description: The solicited administration-site events were erythema, pain and swelling at the injection site.
Time Frame: During the 4-day follow up period after first vaccination (vaccine administered on Day 1)
Population: The analysis was performed on the Exposed Set (ES), which included all participants who received at least 1 dose of the study intervention and for whom solicited administration-site data was available for the specific duration.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 989 | 328 | 329
Participants
  Erythema: number analyzed (Participants) | 989 | 328 | 328
  Erythema | 99 | 38 | 22
  Pain: number analyzed (Participants) | 989 | 328 | 328
  Pain | 595 | 201 | 200
  Swelling: number analyzed (Participants) | 989 | 328 | 328
  Swelling | 75 | 33 | 16

52. Secondary Outcome: Number of Participants With at Least One Solicited Administration-site Event Following Vaccination at Month 12
Description: Month 12 to Month 18 data will be disclosed during final posting. The solicited administration-site events were erythema, pain and swelling at the injection site.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 12)
Reporting Status: Not Posted

53. Secondary Outcome: Number of Participants With at Least One Solicited Administration-site Event Following Vaccination at Month 24
Description: Month 24 data will be disclosed during final posting. The solicited administration-site events were erythema, pain and swelling at the injection site.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 24)
Reporting Status: Not Posted, anticipated posting 2027-05

54. Secondary Outcome: Number of Participants With at Least One Solicited Systemic Event Following Vaccination at Day 1
Description: The solicited systemic events included arthralgia, fatigue, fever (defined as temperature equal to or above 38.0 degree Celsius [°C]), headache and myalgia.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered on Day 1)
Population: The analysis was performed on the ES, which included all participants who received at least 1 dose of the study intervention and for whom solicited systemic data was available for the specific duration.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 989 | 328 | 329
Participants
  Arthralgia | 157 | 49 | 49
  Fatigue | 307 | 100 | 110
  Fever | 13 | 5 | 7
  Headache | 187 | 70 | 79
  Myalgia | 336 | 107 | 109

55. Secondary Outcome: Number of Participants With at Least One Solicited Systemic Event Following Vaccination at Month 12
Description: Month 12 to Month 18 data will be disclosed during final posting. The solicited systemic events included arthralgia, fatigue, fever (defined as temperature equal to or above 38.0°C), headache and myalgia.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 12)
Reporting Status: Not Posted

56. Secondary Outcome: Number of Participants With at Least One Solicited Systemic Event Following Vaccination at Month 24
Description: Month 24 data will be disclosed during final posting. The solicited systemic events included arthralgia, fatigue, fever (defined as temperature equal to or above 38.0 degree Celsius (°C)), headache and myalgia.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 24)
Reporting Status: Not Posted, anticipated posting 2027-05

57. Secondary Outcome: Number of Participants With Any Unsolicited Adverse Events (AEs) Following Vaccination at Day 1
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of study intervention, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study, and/or any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day follow up period after vaccination (vaccine administered on Day 1)
Population: The analysis was performed on the ES, which included all participants who received at least 1 dose of the study intervention and for whom safety data was available for 30 days following vaccination at Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 993 | 329 | 331
Participants | 125 | 45 | 55

58. Secondary Outcome: Number of Participants With Any Unsolicited AEs Following Vaccination at Month 12
Description: Month 12 to Month 18 data will be disclosed during final posting. An unsolicited AE covers any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of study intervention, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study, and/or any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 12)
Reporting Status: Not Posted

59. Secondary Outcome: Number of Participants With Any Unsolicited AEs Following Vaccination at Month 24
Description: Month 24 data will be disclosed during final posting. An unsolicited AE covers any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of study intervention, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study, and/or any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 24)
Reporting Status: Not Posted, anticipated posting 2027-05

60. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) Following Vaccination at Day 1
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study participant.
Time Frame: From first vaccination (Day 1) up to 6 months post-Dose 1 (Month 6)
Population: The analysis was performed on the ES, which included all participants who received at least 1 dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 993 | 329 | 331
Participants | 36 | 16 | 15

61. Secondary Outcome: Number of Participants With SAEs Following Vaccination at Month 12
Description: Month 12 to Month 18 data will be disclosed during final posting. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study participant.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 12)
Reporting Status: Not Posted

62. Secondary Outcome: Number of Participants With SAEs Following Vaccination at Month 24
Description: Month 24 data will be disclosed during final posting. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study participant.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 24)
Reporting Status: Not Posted, anticipated posting 2027-05

63. Secondary Outcome: Number of Participants Reporting Any Potential Immune-mediated Disease (pIMD) Following Vaccination at Day 1
Description: pIMDs are a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From first vaccination (Day 1) up to 6 months post-Dose 1 (Month 6)
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
Number analyzed (Participants) | 993 | 329 | 331
Participants | 0 | 1 | 0

64. Secondary Outcome: Number of Participants Reporting Any pIMD Following Vaccination at Month 12
Description: Month 12 to Month 18 data will be disclosed during final posting. pIMDs are a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 12)
Reporting Status: Not Posted

65. Secondary Outcome: Number of Participants Reporting Any pIMD Following Vaccination at Month 24
Description: Month 24 data will be disclosed during final posting. pIMDs are a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: During the 4-day follow up period after vaccination (vaccine administered at Month 24)
Reporting Status: Not Posted, anticipated posting 2027-05

66. Secondary Outcome: Number of Participants With a Fatal SAE, Related SAE and Related pIMDs
Description: A fatal SAE is any untoward medical occurrence that results in death. A related SAE is an SAE considered to be causally related to the study intervention. A related pIMD is a pIMD considered to be causally related to the study intervention.
  The study is ongoing at the time of the results posting. Results for Months 18 up to study end (Month 36) will be updated during final posting.
Time Frame: From first vaccination (Day 1) up to study end (Month 36)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected from Day 1 to Month 12. Non-serious adverse (Other Adverse events) events were collected within 30 days following first vaccination (vaccine administered at Day 1)
Arm/Group | RSV_annual | RSV_flexible Revaccination | RSV_1dose
All-Cause Mortality (participants affected / at risk) | 3/993 | 1/329 | 3/331
Serious Adverse Events (participants affected / at risk) | 46/993 | 16/329 | 19/331
Other Adverse Events (participants affected / at risk) | 744/993 | 251/329 | 253/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_annual (N=993) | RSV_flexible Revaccination (N=329) | RSV_1dose (N=331)
Coronary artery disease (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Extranodal marginal zone B-cell lymphoma (BALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Iris neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Craniofacial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy in malignant disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chondrolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sacroiliac joint dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 7 (7) | 4 (4) | 5 (5)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_annual (N=993) | RSV_flexible Revaccination (N=329) | RSV_1dose (N=331)
Chills (General disorders) | 6 (6) | 3 (3) | 0 (0)
Injection site pruritus (General disorders) | 8 (8) | 2 (2) | 0 (0)
Fatigue (General disorders) | 307 (308) | 101 (101) | 110 (113)
Asthenia (General disorders) | 2 (2) | 2 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 14 (14) | 6 (6) | 8 (8)
Vaccination site pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 595 (596) | 201 (201) | 200 (201)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site scar (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 77 (77) | 33 (33) | 17 (17)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 162 (167) | 50 (51) | 50 (51)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 337 (339) | 108 (111) | 110 (110)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 192 (198) | 72 (77) | 81 (87)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bursa injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 99 (99) | 38 (38) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT04732871/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT04732871/SAP_001.pdf